CLINICAL TRIAL: NCT02502994
Title: Phase 1 Dose-escalation, Safety / Tolerability and Preliminary Efficacy Study of Intratumoral and Subcutaneous Administration of GEN0101 in Patients With Recurrence of Castration Resistant Prostate Cancer
Brief Title: Phase 1 Study of GEN0101 in Patients With Recurrence of CRPC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norio Nonomura (Other)
Responsible Party: Sponsor-Investigator, Norio Nonomura, Professor, Osaka University
Organization: Osaka University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN0101-JM002
Record Dates: First submitted 2015-05-12; First posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Castration Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Other): Single arm of the castration resistant prostate cancer
  Interventions: Drug: GEN0101

INTERVENTIONS:
Drug: GEN0101

SUMMARY:
This study is designed to evaluate the safety and efficacy of a single injection of GEN0101 in patients with recurrence of castration resistant prostate cancer.

The subjects receive GEN0101 injection 4 times per two weeks (1st intratumoral injection and followed subcutaneous injection) and two weeks of observation as one cycle treatment period. Each subject receive two cycle treatment period.

Low dose group: 30,000m NAU per injection of GEN0101 High dose group: 60,000m NAU per injection of GEN0101 Each group included minimal 3 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients providing a written informed consent by voluntary agreement.
2. Age 20 =< and =<85 years old at the time of informed consent
3. Have a diagnosis of malignant tumor as confirmed by histology or cytology.
4. Have a diagnosis of recurrence of castration resistant prostate cancer and meet the following condition

   * Inapplicable to the standard treatment, ineffective through the criteria of the Prostate Cancer Clinical Trials Working Group (PCWG2) or refuse the standard treatment
   * More than 6 week between the end date of the standard treatment and the registration date when the standard treatment has been ineffective
5. Serum PSA <100 ng/mL at the screening visit
6. Expected survival period is more than 8 weeks after planned start date of investigational product
7. ECOG Performance Status 0 or 1
8. Have an injectable intraprostatic lesion confirmed by histologic examination
9. The marrow function, liver function and the kidney function must be kept as follows at the screening visit (1) leukocyte >= 3,000/mcL (2) neutrophil >=1,500/mcL (3) platelet >=75,000/mcL (4) hemoglobin >=8.0 g/dL. (5) AST =<100 IU/L (6) ALT =<100 IU/L (7) total bilirubin =<2.5 mg/dL (8) serum creatinine =<2.5 mg/dL

Exclusion Criteria:

1. Have multiple brain metastases
2. Positive result of the prick test of GEN0101
3. Have serious complications such as uncontrolled active infection
4. Received systemic chemotherapy, radiotherapy or immunotherapy within 6 weeks before the planned registration date However the hormone therapy except for the estramustine, enzalutamide and abiraterone, bisphosphonate and anti-RANKL antigen antibody is are not included in the systemic chemotherapy.
5. Received another investigational medical product within 4 weeks before the informed concent
6. Had a history of malignancy other than prostate cancer, except for the relapse-free and metastasis-free for more than 5 years after the last treatment at the registration
7. Have an active autoimmune disease
8. Receiving systemic administration of glucocorticosteroid which restrains immunity response, except for the administration for a long period (over 6 months) of the low dose (equivalent to under 10 mg/day oral prednisolone).
9. Had a history of the autologous or homogeneous organ or tissue transplantation (Receiving immunosuppressive medication)
10. PT(%) less than 10% of the lower limit of normal or APTT more than 1.5 times of the upper limit of normal of local reference range at the screening visit
11. Positive result of the hepatitis B surface antigen, HCV antibody or HIV test at the screening visit
12. Inappropriate to be enrolled in this study judged by the investigators

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
DLT (Dose Limiting Toxicity) | 8 weeks
  To determine the appropriate dosing strategy for GEN0101 for castration resistant prostate cancer

SECONDARY OUTCOMES:
Number of participants with tumor shrinkage according to the RECIST. | 8 weeks
Change from baseline in tumor marker (PSA: Prostate Specific Antigen, NSE: Neuron-specific enolase, CEA: Carcinoembryonic Antigen, and CA19-9: Carbohydrate Antigen19-9) at Cycle 1, Week 4 and at Cycle 2, Week 4. | 8 weeks
Change from baseline in prostate histological evaluation at Cycle2, Week2. | 8 weeks
Change from baseline in induction of antitumor immunity (NK cell activity, IL-6 and IFN-gamma) at Cycle1, Week 2 and Week 4 and at Cycle2, Week 2 and Week 4. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Norio Nonomura, MD, Study Chair — Urology, Osaka University Hospital
Locations (1):
- Urology, Osaka University Hospital, Suita, Osaka, Japan